CLINICAL TRIAL: NCT06524297
Title: The Role of a Metaverse Surgical Simulation System in Guiding Incision Site Selection for Uniportal Video-Assisted Thoracoscopic Surgery
Brief Title: The Training of Resident Surgeons in Single-Port Thoracoscopic Surgery Wound Position Selection
Acronym: OpVerse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202407156RINB
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-07

CONDITIONS: Surgical Education
Keywords: Metaverse; Surgical Education; Surgical Simulation; Digital Twin; Mixed Reality; Single-Port Thoracoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metaverse system (Experimental): Residents use the Metaverse system before surgery to simulate wound closure locations on digital twin organs of the patient.
  Interventions: Other: Metaverse system (Patients); Other: Metaverse system (Resident Physician)
- Crontrol group (No Intervention): The control group do not use the Metaverse system.

INTERVENTIONS:
Other: Metaverse system (Patients) — The experimental group will undergo preoperative training using the metaverse surgical simulation system for 15 minutes before selecting the surgical incision site (this refers to residents receiving the assisted training). The trial process requires participants' consent to provide high-resolution CT images as the basis for reconstructing digital twin organs. Except for the intervention training, the surgery, postoperative care, follow-up, and other treatment processes the participants receive will be the same as those for typical patients.
  Arms: Metaverse system
Other: Metaverse system (Resident Physician) — The participants (residents) will receive 15 minutes of preoperative training using the Metaverse surgical simulation system. They will superimpose the digital twin model onto the patient on the operating table and use the CT cross-sectional matching function within the Metaverse system to locate the lesion. The participants (residents) can use the system to repeatedly simulate incision sites and mark planned entry points on the patient by overlaying the virtual model onto the real patient. Except for the intervention training with the system, the subsequent surgery, postoperative care, follow-up, and other treatment processes the patients receive will be the same as usual.
  Arms: Metaverse system

SUMMARY:
the metaverse system applied to the training of wound location selection for singleport thoracoscopic surgery. The experimental design is two groups of 40 computer tomography located superficially less than 2 cm lung nodule patients, one group uses the metaverse system to let resident physicians simulate the wound position on the digital twin organs of each patient, and the other group does not use it. The investigators will evaluate the surgeon's satisfaction with the surgical wound position and urgicalrelated results (such as surgery time, blood loss, etc.). The investigators expect that the system will help improve the appropriateness of resident physicians' choice of wound location for high-difficulty single-port thoracoscopic surgery, help them cross the first threshold necessary to familiarize themselves with the surgery faster, and accelerate learning.

DETAILED DESCRIPTION:
The evolution of single-port thoracoscopic surgery, due to advancements in instrumentation and video technology, has seen a leap in progress since the 2010s.

Today, single-port thoracoscopic surgery has become the mainstream at NTU Thoracic Surgery, capable of performing simple wedge resections or complex pneumonectomies. Single-port thoracoscopic surgery, using only a single wound, aids patients in quickly regaining their preoperative normal life functions, with further reductions in pain. However, its learning curve is steep, with the appropriate choice of wound location being one of the most important thresholds for resident physicians to master this technique. Currently, NTU Surgery and the Media Lab have jointly developed a metaverse surgical simulation platform (OpVerse), creating digital twin organ models through 3D reconstruction software and modeling engines. In mixed reality, including lesion location and anatomical variations, are no different from specific real patients. Users can view and operate CT images and 3D models arbitrarily, mark important structural positions and directions, and measure distances with an XR helmet. The model can also be cross-referenced with CT through cross-sectional positioning. The investigators set up a thoracoscopic simulation lens in the system, superimposing the digital twin model on the patient on the operating table, and using the CT cross-section comparison function in the metaverse system to find the lesion location, resident physicians can repeatedly simulate the wound position through the system, and mark the expected entry wound position on the patient through virtual reality overlay. This project plans to conduct a randomized trial to explore the effectiveness of the metaverse system applied to the training of wound location selection for singleport thoracoscopic surgery. The experimental design is two groups of 40 computer tomography located superficially less than 2 cm lung nodule patients, one group uses the metaverse system to let resident physicians simulate the wound position on the digital twin organs of each patient, and the other group does not use it. The investigators will evaluate the surgeon's satisfaction with the surgical wound position and surgical related results (such as surgery time, blood loss, etc.).

The investigators expect that the system will help improve the appropriateness of resident physicians' choice of wound location for high-difficulty single-port thoracoscopic surgery, help them cross the first threshold necessary to familiarize themselves with the surgery faster, and accelerate learning.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Diagnosed with a lung nodule no larger than 2cm in diameter. The lesion depth must be located within the outer third of the lung.
* Scheduled to undergo computer tomography-guided single-port thoracoscopic wedge resection at National Taiwan University Hospital (NTUH) or National Taiwan Cancer Center (NTUCC).
* Participants who have provided written informed consent for their imaging data to be used by the team to create digital twin models.

Exclusion Criteria:

* Patients with lesions larger than 2 cm.
* Patients not planned for single-port thoracoscopic wedge resection with computed tomography localization.
* Patients who have not provided written consent.
* Members of vulnerable populations.

Inclusion Criteria (Resident Physician):

* Third-year to fifth-year residents in the Department of Thoracic Surgery at National Taiwan University Hospital.

Exclusion Criteria (Resident Physician):

* Residents who are unwilling to participate in the study and decline to sign the consent form.
* Residents with a history of cybersickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Operation time | 24 hours
  Compare the length of operation time between the experimental group (trained using the Metaverse surgical simulation system for 15 minutes pre-operatively) and the control group. This analysis will assess whether pre-operative simulation training reduces operation time for residents.

SECONDARY OUTCOMES:
Satisfaction Questionnaire for Attending Physicians | Through study completion, an average of 1 year.
  To improve the residents selection of wound locations during single-port thoracoscopic surgery, the attending physician will complete a post-operative questionnaire regarding the residents' pre-operative simulation training.

CONTACTS AND LOCATIONS:
Overall Officials: Xu-Heng Chiang, MD, Principal Investigator — Department of Surgery, National Taiwain University Hospital

IPD SHARING:
Plan to Share IPD: No